CLINICAL TRIAL: NCT00635128
Title: Evaluation of GSK Biological's dTpa-IPV Booster Vaccine in Children and Adolescents, 5 Years After Previous dTpa-IPV Boosting.
Brief Title: Safety and Immunogenicity of a Booster Dose of GSK Biological's Boostrix-Polio Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110947
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Results first posted 2017-07-05 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2017-04

CONDITIONS: Poliomyelitis; Diphtheria; Tetanus; Acellular Pertussis
Keywords: Diphtheria; vaccine; DTP; Poliomyelitis; Pertussis; Booster; Tetanus
MeSH Terms: conditions — Poliomyelitis; Diphtheria; Tetanus; Whooping Cough

ARMS (2):
- BOOSTRIX-POLIO GROUP (Experimental): Healthy male or female subjects aged 9 to 13 years, who were given a single booster dose of Boostrix™-Polio vaccine in the dTpa-IPV-001 (711866/001) study, additionally received a single booster dose of the Boostrix™-Polio vaccine, administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Boostrix-Polio
- BOOSTRIX + IPV MÉRIEUX GROUP (Experimental): Healthy male or female subjects aged 9 to 13 years, who were given a single booster dose of Boostrix™ and IPV Mérieux® vaccines in the dTpa-IPV-001 (711866/001) study, additionally received a single booster dose of the Boostrix™-Polio vaccine, administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Boostrix-Polio

INTERVENTIONS:
Biological: Boostrix-Polio — A single booster dose of dTpa-IPV vaccine will be administered to all subjects. IM administration in the deltoid muscle of the non-dominant arm.

SUMMARY:
Subjects aged 9 to 13 years who participated in the 711866/001 study 5 years ago will be evaluated for immune persistence and will receive a combined dTpa-IPV booster dose that will be evaluated in terms of immunogenicity, safety and reactogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they or their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female subject who received a booster vaccination with dTpa-IPV or dTpa + IPV in study 711866/001.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Females of childbearing potential at the time of study entry must have a negative pregnancy test prior to administration of the dose of vaccine and are required to be abstinent or to use adequate contraceptive precautions for one month prior to vaccination. Subjects are required to agree to continue such precautions for two months after vaccination.
* Written informed consent obtained from both parents/ guardians of the subject; assent from the subject himself/herself should also be requested whenever possible.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the booster dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressant or other immune-modifying drugs within six months prior to the booster dose.
* Administration of a vaccine not foreseen by the study protocol within 30 days prior to vaccination, or planned administration during study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Previous booster vaccination against tetanus, diphtheria, pertussis, or poliomyelitis since the booster dose received in study 711866/001.
* History of diphtheria, tetanus, pertussis, or poliomyelitis diseases.
* Any confirmed or suspected immunosuppressive or immunodeficiency condition, based on medical history and physical examination.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Administration of immunoglobulin and/or any blood products within the three months preceding the booster dose or planned administration during the study period.
* Occurrence of transient thrombocytopenia or neurological complications following an earlier immunisation against diphtheria and/or tetanus.
* Occurrence of any of the following adverse events (AEs) after a previous administration of a DTP vaccine: hypersensitivity reaction to any component of the vaccine, encephalopathy of unknown aetiology occurring within 7 days following previous vaccination with pertussis-containing vaccine, fever ≥ 40°C within 48 hours of vaccination not due to another identifiable cause, collapse or shock-like state within 48 hours of vaccination
* Persistent, severe, inconsolable screaming or crying lasting >3 hours occurring within 48 hours of receipt of a previous dose of DTP vaccine convulsions with or without fever, occurring within 3 days of vaccination.
* Acute disease at the time of enrolment.
* Pregnant or lactating female.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 415 (Actual)
Dates: Start 2008-02-01 (Actual); Primary Completion 2008-07-08 (Actual); Study Completion 2008-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (32):
- Germany (32):
  - GSK Investigational Site, Ettenheim, Baden-Wurttemberg
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Oberkirch, Baden-Wurttemberg
  - GSK Investigational Site, Offenburg, Baden-Wurttemberg
  - GSK Investigational Site, Cham, Bavaria
  - GSK Investigational Site, Kaufering, Bavaria
  - GSK Investigational Site, Landshut, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Olching, Bavaria
  - GSK Investigational Site, Weilheim, Bavaria
  - GSK Investigational Site, Eschwege, Hesse
  - GSK Investigational Site, Koenigstein, Hesse
  - GSK Investigational Site, Salzgitter, Lower Saxony
  - GSK Investigational Site, Wolfenbüttel, Lower Saxony
  - GSK Investigational Site, Erkrath, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Gütersloh, North Rhine-Westphalia
  - GSK Investigational Site, Heiligenhaus, North Rhine-Westphalia
  - GSK Investigational Site, Kleve-Materborn, North Rhine-Westphalia
  - GSK Investigational Site, Krefeld, North Rhine-Westphalia
  - GSK Investigational Site, Löhne, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Willich, North Rhine-Westphalia
  - GSK Investigational Site, Bad Kreuznach, Rhineland-Palatinate
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Worms, Rhineland-Palatinate
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Brunsbüttel, Schleswig-Holstein
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Berlin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Knuf M et al. The repeated administration of a reduced antigen content diphtheria, tetanus, acellular pertussis and poliomyelitis vaccine (dTpa-IPV; BoostrixTM IPV) in adolescents. Abstract presented at IDSA. Philadelphia, USA, 29 October- 1 November 2009.
- [Background] Knuf M, Baine Y, Bianco V, Boutriau D, Miller JM. Antibody persistence and immune memory 15 months after priming with an investigational tetravalent meningococcal tetanus toxoid conjugate vaccine (MenACWY-TT) in toddlers and young children. Hum Vaccin Immunother. 2012 Jul;8(7):866-72. doi: 10.4161/hv.20229. Epub 2012 Apr 9. PMID 22485049
- [Background] Mertsola J et al. The safety of repeated administration of Boostrix™, a reduced-antigen-content dTpa booster. Abstract presented at Excellence In Paediatrics (EIP). Florence, Italy, 3-6 December 2009.
- [Background] Mertsola J et al. The safety of repeated administration of reduced-antigen-content dTpa boosters. Abstract presented at WSPID-6th World Congress. Buenos Aires, Argentina, 19-22 November 2009.
- [Derived] Knuf M, Vetter V, Celzo F, Ramakrishnan G, Van Der Meeren O, Jacquet JM. Repeated administration of a reduced-antigen-content diphtheria-tetanus-acellular pertussis and poliomyelitis vaccine (dTpa-IPV; Boostrix IPV). Hum Vaccin. 2010 Jul;6(7):554-61. doi: 10.4161/hv.6.7.11760. PMID 20448468
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 110947 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110947 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110947 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110947 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110947 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110947 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110947 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Boostrix-Polio Group: Healthy male or female subjects aged 9 to 13 years, who were given a single booster dose of Boostrix-Polio vaccine in the dTpa-IPV-001 (711866/001) study, additionally received a single booster dose of the Boostrix-Polio vaccine, administered intramuscularly in the deltoid region of the non-dominant arm.
- Boostrix + IPV Mérieux Group: Healthy male or female subjects aged 9 to 13 years, who were given a single booster dose of Boostrix and IPV Mérieux® vaccines in the dTpa-IPV-001 (711866/001) study, additionally received a single booster dose of the Boostrix-Polio vaccine, administered intramuscularly in the deltoid region of the non-dominant arm.
Period: Overall Study
Arm/Group | Boostrix-Polio Group | Boostrix + IPV Mérieux Group
Started | 351 | 64
Completed | 351 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Boostrix-Polio Group | Boostrix + IPV Mérieux Group | Total
Number analyzed (Participants) | 351 | 64 | 415
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.4 (0.97) | 11.3 (0.72) | 11.38 (0.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169 | 32 | 201
  Male | 182 | 32 | 214
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White-Caucasian/European heritage | 347 | 63 | 410
  White-Arabic/North African heritage | 4 | 0 | 4
  Not specified | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Grade 3 Pain: Pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: During the 4-day (Days 0-3) follow-up period after booster vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix-Polio Group | Boostrix + IPV Mérieux Group
Number analyzed (Participants) | 351 | 64
Participants
  Grade 3 Pain | 14 | 3
  Grade 3 Redness (mm) | 14 | 5
  Grade 3 Swelling (mm) | 10 | 5

2. Secondary Outcome: Number of Subjects With Any Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 4-day (Days 0-3) follow-up period after booster vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix-Polio Group | Boostrix + IPV Mérieux Group
Number analyzed (Participants) | 351 | 64
Participants
  Any Pain | 257 | 45
  Any Redness | 169 | 26
  Any Swelling | 141 | 22

3. Secondary Outcome: Number of Subjects With Any Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal, headache and temperature [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade and relationship to vaccination.
Time Frame: During the 4-day (Days 0-3) follow-up period after booster vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects for whom data were available and who had the symptoms sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix-Polio Group | Boostrix + IPV Mérieux Group
Number analyzed (Participants) | 351 | 63
Participants
  Any Fatigue | 87 | 14
  Any Gastrointestinal | 41 | 4
  Any Headache | 76 | 12
  Any Temperature | 14 | 0

4. Secondary Outcome: Number of Subjects With Anti-diphtheria (Anti-D) and Anti-tetanus (Anti-T) Toxoids
Description: Anti-D and anti-T antibody concnetration greater than or equal to (≥) 0.1 international units per milliliter (IU/mL) and ≥ 1 IU/mL have been assessed by enzyme-linked immunosorbent assay (ELISA). Pre-vaccination sera with ELISA concentrations < 0.1 IU/mL were tested for neutralising antibodies using a Vero-cell neutralisation assay with a 0.016 IU/mL cut-off.
Time Frame: Prior to (Month 0) and one month after (Month 1) booster vaccination
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects vaccinated with a booster dose of Boostrix™-Polio vaccine in this current study (110947), for whom immunogenicity data and assay results for antibodies against at least one study vaccine antigen component were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix-Polio Group | Boostrix + IPV Mérieux Group
Number analyzed (Participants) | 336 | 62
Participants
  Anti-D ≥ 0.1 IU/mL, M0: number analyzed (Participants) | 334 | 62
  Anti-D ≥ 0.1 IU/mL, M0 | 298 | 53
  Anti-D ≥ 0.1 IU/mL, M1 | 336 | 62
  Anti-D ≥ 1 IU/mL, M0: number analyzed (Participants) | 334 | 62
  Anti-D ≥ 1 IU/mL, M0 | 91 | 13
  Anti-D ≥ 1 IU/mL, M1 | 308 | 55
  Anti-T ≥ 0.1 IU/mL, M0: number analyzed (Participants) | 335 | 62
  Anti-T ≥ 0.1 IU/mL, M0 | 330 | 61
  Anti-T ≥ 0.1 IU/mL, M1 | 336 | 62
  Anti-T ≥ 1 IU/mL, M0: number analyzed (Participants) | 335 | 62
  Anti-T ≥ 1 IU/mL, M0 | 181 | 35
  Anti-T ≥ 1 IU/mL, M1 | 335 | 61

5. Secondary Outcome: Anti-D and Anti-T Antibody Concentrations
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in international units per milliliter (IU/mL).
Time Frame: Prior to (Month 0) and one month after (Month 1) booster vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix-Polio Group | Boostrix + IPV Mérieux Group
Number analyzed (Participants) | 336 | 62
IU/mL
  Anti-D, M0: number analyzed (Participants) | 334 | 62
  Anti-D, M0 | 0.51 [0.429 to 0.608] | 0.446 [0.305 to 0.651]
  Anti-D, M1 | 4.784 [4.302 to 5.32] | 4.153 [3.089 to 5.585]
  Anti-T, M0: number analyzed (Participants) | 335 | 62
  Anti-T, M0 | 1.197 [1.045 to 1.37] | 1.067 [0.797 to 1.429]
  Anti-T, M1 | 11.81 [11.011 to 12.667] | 9.518 [7.879 to 11.498]

6. Secondary Outcome: Number of Seropositive Subjects for Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN)
Description: A seropositive subject was defined as a subject with anti-PT, anti-FHA and anti-PRN antibody concentrations ≥ 5 ELISA unit per milliliter (EL.U/ml).
Time Frame: Prior to (Month 0) and one month after (Month 1) booster vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix-Polio Group | Boostrix + IPV Mérieux Group
Number analyzed (Participants) | 336 | 62
Participants
  Anti-PT, M0: number analyzed (Participants) | 330 | 62
  Anti-PT, M0 | 134 | 21
  Anti-PT, M1: number analyzed (Participants) | 335 | 62
  Anti-PT, M1 | 334 | 59
  Anti-FHA, M0: number analyzed (Participants) | 333 | 60
  Anti-FHA, M0 | 332 | 60
  Anti-FHA, M1: number analyzed (Participants) | 336 | 61
  Anti-FHA, M1 | 336 | 61
  Anti-PRN, M0: number analyzed (Participants) | 335 | 62
  Anti-PRN, M0 | 325 | 57
  Anti-PRN, M1 | 336 | 62

7. Secondary Outcome: Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations
Description: Antibodies concentrations were presented as geometric mean concentrations (GMCs), expressed in EL.U/mL.
Time Frame: Prior to (Month 0) and one month after (Month 1) booster vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Boostrix-Polio Group | Boostrix + IPV Mérieux Group
Number analyzed (Participants) | 336 | 62
EL.U/mL
  Anti-PT, M0: number analyzed (Participants) | 330 | 62
  Anti-PT, M0 | 5.2 [4.7 to 5.9] | 4.5 [3.6 to 5.6]
  Anti-PT, M1: number analyzed (Participants) | 335 | 62
  Anti-PT, M1 | 41.6 [38.1 to 45.3] | 32 [24.5 to 41.9]
  Anti-FHA, M0: number analyzed (Participants) | 333 | 60
  Anti-FHA, M0 | 69.8 [62.1 to 78.4] | 70.1 [52.5 to 93.5]
  Anti-FHA, M1: number analyzed (Participants) | 336 | 61
  Anti-FHA, M1 | 662.7 [613.2 to 716.1] | 733.9 [610.4 to 882.5]
  Anti-PRN, M0: number analyzed (Participants) | 335 | 62
  Anti-PRN, M0 | 46.8 [41.5 to 52.8] | 41.1 [30 to 56.2]
  Anti-PRN, M1 | 570.8 [527.4 to 617.7] | 460.4 [353.3 to 600]

8. Secondary Outcome: Number of Seroprotected Subjects Against Polio Type 1, 2 and 3 Antigens
Description: A seroprotected subject was defined as a subject with anti-Polio type 1, 2 and 3 antibody titers ≥ the value of 8.
Time Frame: Prior to (Month 0) and one month after (Month 1) booster vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix-Polio Group | Boostrix + IPV Mérieux Group
Number analyzed (Participants) | 335 | 62
Participants
  Anti-polio 1, M0: number analyzed (Participants) | 333 | 62
  Anti-polio 1, M0 | 329 | 60
  Anti-polio 1, M1 | 335 | 62
  Anti-polio 2, M0: number analyzed (Participants) | 334 | 62
  Anti-polio 2, M0 | 333 | 62
  Anti-polio 2, M1 | 335 | 62
  Anti-polio 3, M0: number analyzed (Participants) | 334 | 62
  Anti-polio 3, M0 | 324 | 60
  Anti-polio 3, M1: number analyzed (Participants) | 333 | 62
  Anti-polio 3, M1 | 333 | 62

9. Secondary Outcome: Anti-Polio 1, 2 and 3 Antibody Titers
Description: Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: Prior to (Month 0) and one month after (Month 1) booster vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Boostrix-Polio Group | Boostrix + IPV Mérieux Group
Number analyzed (Participants) | 335 | 62
Titers
  Anti-polio 1, M0: number analyzed (Participants) | 333 | 62
  Anti-polio 1, M0 | 138.7 [123 to 156.4] | 128.9 [96.1 to 172.7]
  Anti-polio 1, M1 | 1359.6 [1213.4 to 1523.3] | 1088.9 [866.5 to 1368.4]
  Anti-polio 2, M0: number analyzed (Participants) | 334 | 62
  Anti-polio 2, M0 | 166.3 [149.5 to 185] | 179.2 [142.9 to 224.7]
  Anti-polio 2, M1 | 1629.4 [1475.2 to 1799.7] | 1309.5 [1035.2 to 1656.3]
  Anti-polio 3, M0: number analyzed (Participants) | 334 | 62
  Anti-polio 3, M0 | 117.2 [102.8 to 133.5] | 118.4 [83.4 to 168]
  Anti-polio 3, M1: number analyzed (Participants) | 333 | 62
  Anti-polio 3, M1 | 1882.4 [1687.9 to 2099.3] | 1712.5 [1329.2 to 2206.3]

10. Secondary Outcome: Number of Subjects With Booster Response to Anti-PT, Anti-FHA and Anti-PRN
Description: Booster vaccine response was defined as appearance of antibodies in subjects who were seronegative at the pre-vaccination time point (i.e. with concentrations < 5 EL.U/mL) or at least 2-fold increase of pre-vaccination antibody concentrations in subjects who were seropositive at the pre-vaccination time point (i.e. with concentrations < 5 EL.U/mL).
Time Frame: One month after booster vaccination (At Month 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix-Polio Group | Boostrix + IPV Mérieux Group
Number analyzed (Participants) | 335 | 62
Participants
  Anti-PT: number analyzed (Participants) | 330 | 62
  Anti-PT | 308 | 56
  Anti-FHA: number analyzed (Participants) | 333 | 60
  Anti-FHA | 311 | 56
  Anti-PRN | 319 | 61

11. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: AEs results are presented for all subjects. An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0-30) follow-up period after booster vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix-Polio Group | Boostrix + IPV Mérieux Group
Number analyzed (Participants) | 351 | 64
Participants | 47 | 17

12. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Assessed SAEs include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire booster period (Month 0 to Month 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix-Polio Group | Boostrix + IPV Mérieux Group
Number analyzed (Participants) | 351 | 64
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms during the 4-day (Days 0-3) post-booster period; AEs during the 31-day (Days 0-30) post-booster period; SAEs following booster vaccination (up to Month 1).
Arm/Group | Boostrix-Polio Group | Boostrix + IPV Mérieux Group
All-Cause Mortality (participants affected / at risk) | 0/351 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/351 | 0/64
Other Adverse Events (participants affected / at risk) | 281/351 | 51/64
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Boostrix-Polio Group (N=351) | Boostrix + IPV Mérieux Group (N=64)
Pain (General disorders) | 257 | 45
Redness (mm) (General disorders) | 169 | 26
Swelling (mm) (General disorders) | 141 | 22
Fatigue (General disorders) | 87 | 14/63 — This solicited general symptom was collected only from subjects with their symptom sheets completed.
Gastrointestinal symptoms (General disorders) | 41 | 4/63 — This solicited general symptom was collected only from subjects with their symptom sheets completed.
Headache (General disorders) | 76 | 12/63 — This solicited general symptom was collected only from subjects with their symptom sheets completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.